CLINICAL TRIAL: NCT04854642
Title: Influence of Food on the Oral Bioavailability of Ladarixin 200 mg Capsule in Healthy Volunteers of Both Sexes. A Single Dose (400 mg), Randomized, Open Label, Two-Way Crossover Study
Brief Title: A Single Dose Study About the Influence of Food on the Oral Bioavailability of Ladarixin Capsule in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LDX0219
Record Dates: First submitted 2021-04-15; First posted 2021-04-22 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: no Condition
MeSH Terms: interventions — 2'-((4'-trifluoromethanesulfonyloxy)phenyl)-N-methanesulfonylpropionamide

STUDY DESIGN:
Masking Description: This is an open-label trial. No masking procedure will be applied since an open-label design was considered adequate for evaluating objective measures such as pharmacokinetic parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T - R (fed then fasting condition) (Experimental): Subjects were assigned to the sequence of treatments TR to receive Ladarixin in fed conditions (T treatment) during period 1 and in fasting conditions (R treatment) in period 2.
  Interventions: Drug: Ladarixin
- R - T (fasting then fed condition) (Experimental): Subjects were assigned to the sequence of treatments RT to receive Ladarixin ini fasting conditions (R treatment) in period 1 and in fed conditions (T treatment) during period 2.
  Interventions: Drug: Ladarixin

INTERVENTIONS:
Drug: Ladarixin — A single oral dose of 400 mg of ladarixin (two 200 mg capsules) was administered to healthy male and female volunteers under fed (Test treatment) and fasting (Reference treatment) conditions in two consecutive study periods, according to a two-way crossover design, with a wash-out interval of at least 14 days between the two administrations.
  Other Names: LDX

SUMMARY:
Primary objective:

- to investigate the effect of food on the bioavailability of DF 2156Y after single dose administration of 400 mg of ladarixin to healthy male and female volunteers under fed and fasting conditions.

Secondary objectives:

* to investigate the effect of gender on the bioavailability of DF 2156Y and its metabolites (DF 2108Y and DF 2227Y) after single dose administration of 400 mg of ladarixin to healthy male and female volunteers
* to evaluate safety and tolerability of a single dose administration of ladarixin 400 mg to healthy male and female volunteers.

DETAILED DESCRIPTION:
This is a Single center, single dose, open label, randomized, two-way, crossover, food effect on bioavailability study.

More precisely, a single oral dose of 400 mg of ladarixin (two 200 mg capsules) was administered to healthy male and female volunteers under fed (Test treatment) and fasting (Reference treatment) conditions in two consecutive study periods, according to a two-way crossover design, with a wash-out interval of at least 14 days between the two administrations.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: men/women, 18-55 years old inclusive
3. Body Mass Index: 18.5-30 kg/m2 inclusive
4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, pulse rate 50-90 bpm and body temperature 35.5-37.5° C, measured after 5 min at rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
6. Contraception and fertility (women only): women of child-bearing potential must not wish to get pregnant within 30 days after the end of the study and must be using at least one of the following reliable methods of contraception:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit until 30 days after final visit
   2. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit until 30 days after final visit
   3. A male sexual partner who agrees to use a male condom with spermicide until 30 days after final visit
   4. A sterile sexual partner Women participants of non-childbearing potential or in post-menopausal status for at least one year will be admitted. For all women, pregnancy test result must be negative at screening and day -1.

Exclusion Criteria:

1. Electrocardiogram (ECG) 12-leads (supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
4. Allergy: ascertained or presumptive hypersensitivity to the active principles (ladarixin or derivatives) and/or formulations' ingredients; known hypersensitivity to non-steroidal anti-inflammatory drugs (NSAIDs); history of hypersensitivity to drugs (in particular methanesulfonyl propanamide) or allergic reactions in general, which the Investigator considers may affect the outcome of the study
5. Diseases: hypoalbuminemia or significant history of renal, hepatic, gastrointestinal, respiratory, skin, hematological, endocrine, neurological or cardiovascular diseases that may interfere with the aim of the study
6. Medications: medications, including over the counter drugs (in particular nonsteroidal anti-inflammatory drugs), herbal remedies and food supplements taken 14 days before the start of the study (in any case at least 5 times the half-life of the drug or a minimum of 14 days, whichever is longer), with the exception of paracetamol. Hormonal contraceptives and hormonal replacement therapy for women will be allowed.
7. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
8. Blood donation: blood donations for 3 months before this study
9. Drug, alcohol, caffeine, tobacco: history of drug, alcohol (>1 drink/day for women and >2 drinks/day for men, defined according to the USDA Dietary Guidelines 2015-2020), caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes/day)
10. SARS-COV2 test: positive SARS-COV2 test on day -3 or -2 of each study period
11. Virology: positive Hepatitis B (HBs antigen), Hepatitis C (HCV antibodies), HIV 1/2 (HIV Ag/Ab combo) at screening.
12. Drug test: positive result at the drug test at screening or day -1 of each study period
13. Alcohol test: positive alcohol breath test at screening or day -1 of each study period
14. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians; vegans
15. Pregnancy (women only): positive or missing pregnancy test at screening or day -1 of each study period, pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — CROSS Research S.A., I Unit,
Locations (1):
- CROSS Research S.A., I Unit, Arzo, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-six (36) subjects were enrolled in the study, as planned, and 32 of them completed the study as per protocol.
Period: Overall Study
Arm/Group | T - R (Fed Then Fasting Condition) | R - T (Fasting Then Fed Condition)
Started | 18 | 18
Safety Set | 18 | 18
PK Set 1 | 18 | 18
PK Set 2 | 18 | 18
Completed | 17 | 15
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled set: all enrolled subjects. This analysis set was used for demographic, baseline and background characteristics
Groups:
- Enrolled and Safety Set, PK Set 1 and PK Set 2: Demographics are reported for the "enrolled set" (N=36), which has the same number of participants of the "safety set", the "PK set 1", and the "PK set 2".
Arm/Group | Enrolled and Safety Set, PK Set 1 and PK Set 2
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 36

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Plasma DF 2156Y
Description: PK parameters were assessed after single dose administration of 400 mg of ladarixin under fed and fasting conditions.
  Cmax = maximum plasma concentration
Time Frame: At day 1 (15 min, 30 min, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hours postdose); at days 2 and 3 (24, 30, 36, 48, 54 and 60 hours post-dose); at day 4 (72 hours post-dose)
Population: PK set 1: all subjects randomised who fulfilled the study protocol requirements in terms of IMP intake and had evaluable PK data readouts for DF 2156Y with no major deviations that could affect the PK results. This analysis set was used for the statistical analysis of the PK results for DF 2156Y.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Ladarixin Fed (T): Ladarixin - Fed Condition: A single oral dose of 400 mg of ladarixin (two 200 mg capsules) was administered to healthy male and female volunteers under fed (Test treatment) condition.
- Ladarixin Fasting (R): Ladarixin - Fasting condition: A single oral dose of 400 mg of ladarixin (two 200 mg capsules) was administered to healthy male and female volunteers under fasting (Reference treatment) condition.
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
μg/mL | 67.345 (11.426) | 95.982 (14.257)
Statistical Analysis 1: Comparison: Ladarixin Fed (T) vs Ladarixin Fasting (R); Test type: Other; p < 0.0001, ANOVA; Least square mean difference = 71.62, 90% CI 2-sided [68.13 to 75.29]

2. Primary Outcome: AUC0-t of Plasma DF 2156Y
Description: PK parameters were assessed after single dose administration of 400 mg of ladarixin under fed and fasting conditions.
  AUC0-t = area under the concentration-time curve (AUC) from zero to the last quantifiable concentrations
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
h*μg/mL | 1422.500 (362.265) | 1564.189 (364.099)
Statistical Analysis 1: Comparison: Ladarixin Fed (T) vs Ladarixin Fasting (R); Test type: Other; p = 0.0170, ANOVA; Least square mean difference = 90.93, 90% CI 2-sided [85.30 to 96.93]

3. Secondary Outcome: AUC0-∞ of Plasma DF 2156Y
Description: PK parameters were assessed after single dose administration of 400 mg of ladarixin under fed and fasting conditions:
  AUC0-∞ = area under the concentration-time curve (AUC) from zero to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
h*μg/mL | 1533.432 (442.119) | 1677.749 (434.421)
Statistical Analysis 1: Comparison: Ladarixin Fed (T) vs Ladarixin Fasting (R); Test type: Other; p = 0.0213, ANOVA; Least square mean difference = 90.90, 90% CI 2-sided [85.04 to 97.16]

4. Secondary Outcome: Tmax of Plasma DF 2156Y
Description: PK parameters were assessed after single dose administration of 400 mg of ladarixin under fed and fasting conditions.
  tmax = time to maximum plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
h | 5.485 (0.939) | 1.914 (1.197)
Statistical Analysis 1: Comparison: Ladarixin Fed (T) vs Ladarixin Fasting (R); Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: t1/2 of Plasma DF 2156Y
Description: PK parameters were assessed after single dose administration of 400 mg of ladarixin under fed and fasting conditions.
  t1/2 = half life, is the time required for a quantity to reduce to half of its initial value
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
h | 16.918 (5.797) | 17.087 (5.349)

6. Secondary Outcome: Lambda-zeta of Plasma DF 2156Y
Description: PK parameters were assessed after single dose administration of 400 mg of ladarixin under fed and fasting conditions.
  lambda-zeta is the Individual estimate of the terminal elimination rate constant, calculated using log-linear regression of the terminal portions of the plasma concentration-versus-time curves
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
1/h | 0.046 (0.015) | 0.045 (0.015)

7. Secondary Outcome: Frel of Plasma DF 2156Y
Description: PK parameters were assessed after single dose administration of 400 mg of ladarixin under fed and fasting conditions.
  Frel: Relative bioavailability, calculated as ratio AUC0-t (T)/ AUC0-t (R) (multiplicated by 100)
Time Frame: as for outcome 1
Population: PK sets 1 and 2 : PK set 1: all subjects randomised who fulfilled the study protocol requirements in terms of IMP intake and had evaluable PK data readouts for DF 2156Y with no major deviations that could affect the PK results.
  PK set 2: all subjects randomised who fulfilled the study protocol requirements in terms of IMP intake and had evaluable PK data readouts for DF 2108Y and DF 2227Y, with no major deviations that could affect the PK results.
Measure: Mean (Standard Deviation); unit: percentage of bioavailability
Groups:
- Enrolled and Safety Set, PK Set 1 and PK Set 2: Demographics are reported for the "enrolled set" (N=36); which has the same number of participants of the "safety set", the "PK set 1" and the "PK set 2"
Arm/Group | Enrolled and Safety Set, PK Set 1 and PK Set 2
Number analyzed (Participants) | 32
percentage of bioavailability | 93.721 (21.605)

8. Secondary Outcome: Cmax of Plasma DF 2108Y (DF 2156Y Metabolite)
Description: PK parameters were assessed after single dose of 400 mg of ladarixin under fed and fasting conditions.
  Cmax = maximum plasma concentration
Time Frame: as for outcome 1
Population: PK set 2: all subjects randomised who fulfilled the study protocol requirements in terms of IMP intake and had evaluable PK data readouts for DF 2108Y and DF 2227Y, with no major deviations that could affect the PK results. This analysis set was used for the statistical analysis of the PK results for DF 2108Y and DF 2227Y.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
μg/mL | 0.940 (0.292) | 0.972 (0.210)

9. Secondary Outcome: AUC0-t of Plasma DF 2108Y (DF 2156Y Metabolite)
Description: PK parameters were assessed after single dose of 400 mg of ladarixin under fed and fasting conditions.
  AUC0-t = area under the concentration-time curve (AUC) from zero to the last quantifiable concentrations
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: (h*μg/mL
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
(h*μg/mL | 47.013 (13.822) | 50.462 (11.636)

10. Secondary Outcome: AUC0-∞ of Plasma DF 2108Y (DF 2156Y Metabolite)
Description: PK parameters were assessed after single dose of 400 mg of ladarixin under fed and fasting conditions.
  AUC0-∞ = area under the concentration-time curve (AUC) from zero to infinity
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
h*μg/mL | 78.549 (48.921) | 77.220 (29.818)

11. Secondary Outcome: Tmax of Plasma DF 2108Y (DF 2156Y Metabolite)
Description: PK parameters were assessed after single dose of 400 mg of ladarixin under fed and fasting conditions.
  tmax = time to maximum plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
h | 28.364 (5.667) | 24.343 (9.474)

12. Secondary Outcome: t1/2 of Plasma DF 2108Y (DF 2156Y Metabolite)
Description: PK parameters were assessed after single dose of 400 mg of ladarixin under fed and fasting conditions.
  t1/2 = half life, is the time required for a quantity to reduce to half of its initial value
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
h | 40.637 (28.192) | 36.444 (16.315)

13. Secondary Outcome: Lambda-zeta of Plasma DF2108Y (DF 2156Y Metabolite)
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
1/h | 0.022 (0.010) | 0.023 (0.010)

14. Secondary Outcome: Frel of Plasma DF2108Y (DF 2156Y Metabolite)
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of bioavailability
Arm/Group | Enrolled and Safety Set, PK Set 1 and PK Set 2
Number analyzed (Participants) | 32
percentage of bioavailability | 95.569 (20.352)

15. Secondary Outcome: Cmax of Plasma DF2227Y (DF 2156Y Metabolite)
Description: as for outcome 8
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
μg/mL | 0.882 (0.195) | 0.964 (0.192)

16. Secondary Outcome: AUC0-t of Plasma DF2227Y (DF 2156Y Metabolite)
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
h*μg/mL | 52.928 (10.877) | 58.465 (10.884)

17. Secondary Outcome: Tmax of Plasma DF2227Y (DF 2156Y Metabolite)
Description: as for outcome 11
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
Number analyzed (Participants) | 33 | 35
hours | 36.606 (19.349) | 31.657 (23.849)

18. Secondary Outcome: Frel of Plasma DF222Y (DF 2156Y Metabolite)
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of bioavailability
Arm/Group | Enrolled and Safety Set, PK Set 1 and PK Set 2
Number analyzed (Participants) | 32
percentage of bioavailability | 92.745 (13.340)

ADVERSE EVENTS:
Time Frame: Throughout the study, from screening to final visit /ETV (at day 4 of period 2 or early termination up to 22 days)
Description: The TEAE were calculated based on the safety set. The Safety set consists of all subjects who received at least one dose of study treatments. This analysis set was used for the safety and tolerability analyses.
Groups:
- Ladarixin Fed (T): Ladarixin - Fed Conditions: A single oral dose of 400 mg of ladarixin (two 200 mg capsules) was administered to healthy male and female volunteers under fed (Test treatment) conditions.
- Ladarixin Fasting (R): Ladarixin - Fasting conditions: A single oral dose of 400 mg of ladarixin (two 200 mg capsules) was administered to healthy male and female volunteers under fasting (Reference treatment) conditions.
Arm/Group | Ladarixin Fed (T) | Ladarixin Fasting (R)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 4/33 | 4/35
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ladarixin Fed (T) (N=33) | Ladarixin Fasting (R) (N=35)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations and Caveats not specified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT04854642/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04854642/SAP_001.pdf